CLINICAL TRIAL: NCT04159194
Title: Performance and Physiological Analysis of Overtime in Soccer: Implications for Recovery and Training
Brief Title: Analysis of Overtime in Soccer
Acronym: SOCCER-120
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SOCCER-OVERTIME-UTH 2019
Record Dates: First submitted 2019-09-10; First posted 2019-11-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2019-09

CONDITIONS: Metabolic Stress
Keywords: soccer; overtime; performance; recovery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal CHO (Active Comparator)
  Interventions: Other: Control Diet
- High CHO (Experimental)
  Interventions: Other: Experimental Diet

INTERVENTIONS:
Other: Control Diet — Players during the control trial will be instructed to maintain their normal food intake (~55% CHO) and the type and amount of ingested food will be recorded.
  Arms: Normal CHO
Other: Experimental Diet — The experimental diet will be administered by the investigators after M1, daily for the next 48 hours (three main meals, i.e. breakfast, lunch, and dinner, and snacks such as energy bars and raisins), and before M2 (breakfast and lunch)
  Arms: High CHO

SUMMARY:
A randomized, two-trial (placebo vs. supplement consumption), cross-over, double-blind, repeated measures design will be applied to study i) the performance, metabolic and inflammatory overload of overtime in soccer and ii) how carbohydrate supplementation affects recovery following a football match with overtime. The study will be performed during a brake of the in-season period to mimic a real life setting. A 10-day washout period will be utilized between trials.

DETAILED DESCRIPTION:
Initially and before the familiarization period, measurement of descriptive variables will be performed: body composition, maximal oxygen consumption, football-specific endurance via YO-YO IE2 and IR2, technical performance, daily diet intake, resting metabolic rate (canopy method), and daily physical activity (IPAQ questionnaire). At this time, volunteers (of equal technical, tactical and physical potential) will be randomly assigned (equally representing all field positions) to two teams.

A 7-day familiarization period will be applied initially during which participants will be accustomed with research procedures, match tactics, and diet (a standard diet will be given based on their dietary analysis, RMR measurement and daily energy expenditure). During this adaptive period, volunteers will participated in light training aimed at developing team cohesion.

Thereafter, the two experimental trials will take place. Each trial will include administration of either a high carbohydrate diet (CHO trial) or standard diet (control trial) and they will be carried out in a random order for each participant. Each trial will included two 120-min matches (M1 and M2) performed 3 days apart according to UEFA official schedules for National teams' tournaments. On match days, volunteers will participate only in morning testing sessions but not practice. Prior to each game, a standard breakfast and meal will be consumed. During each match, players will be allowed to drink only water ad libitum and their water intake will be recorded. Sweat loss during the match will be determined by measuring players' body mass wearing dry shorts immediately before the match, at half time, immediately after the match and immediately after each half of the overtime. Two practice sessions will take place on days 1 and 2 between M1 and M2 designed according to the training model routinely adapted by national football teams during the UEFA EURO tournament. Matches will be organized according to official UEFA regulations. Field activity during matches and practices will be recorded using high time-resolution GPS instrumentation and heart rate monitoring. Following M1 and for the next 3 days until M2, participants will receive either carbohydrate or placebo. Diet intake will be monitored daily throughout the study.

Performance assessments will be performed post-matches and daily between matches.

Blood samples will be collected at baseline as well as at 90 and 120 min of each match and before M2.

Muscle biopsies will be collected at baseline as well as at 90 and 120 min of M1 and before M2.

ELIGIBILITY:
Inclusion Criteria:

* competitive level for ≥4 years (≥5 training sessions/week, ≥1 match/week)
* no recent history of febrile illness, muscle lesions, lower limb trauma, and metabolic diseases
* no use of ergogenic supplements and medication (for ≥6 prior to the study)
* non-smokers

Exclusion Criteria:

* recent history of febrile illness, muscle lesions, lower limb trauma, and metabolic diseases
* use of ergogenic supplements and medication (for ≥6 prior to the study)
* smoking
* competitive level for < 4 years

Ages: 20 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Measurement of countermovement jump height | Change from baseline to 90 minutes and 120 minutes of the game.
Measurement of maximal sprinting speed over 10 meters | Change from baseline to 90 minutes and 120 minutes of the game.
  10-m sprinting speed will be assessed on the soccer field by utilizing light cells
Measurement of maximal sprinting speed over 30 meters | Change from baseline to 90 minutes and 120 minutes of the game.
  30-m sprinting speed will be assessed on the soccer field by utilizing light cells
Measurement of the capacity to perform repeated sprints | Change from baseline to 90 minutes and 120 minutes of the game.
  5 x 30m repeated maximal sprints will be performed with 30 sec rest in between. Speed will be recorded by utilizing light cells.
Measurement of isometric maximal voluntary contraction | At baseline
  Isometric maximal voluntary contraction will be assessed on an isokinetic dynamometer
Measurement of total protein content | Change from baseline to 90 minutes and 120 minutes of the game.
  Total protein content will be assessed on muscle biopsy samples
Measurement of muscle glycogen content | Change from baseline to 90 minutes and 120 minutes of the game.
  Muscle glycogen content will be assessed on muscle biopsy samples
Measurement of muscle phosphocreatine content | Change from baseline to 90 minutes and 120 minutes of the game.
  Muscle phosphocreatine levels will be assessed on muscle biopsy samples
Measurement of muscle lactate concentration | Change from baseline to 90 minutes and 120 minutes of the game.
  Muscle lactate concentration will be assessed on muscle biopsy samples
Measurement of Na+ - K+ ATPase levels | Change from baseline to 90 minutes and 120 minutes of the game.
  Muscle Na+ - K+ ATPase levels will be assessed on muscle biopsy samples
Measurement of creatine kinase activity | Change from baseline to 90 minutes and 120 minutes of the game.
  Creatine kinase activity will be measured on blood samples
Measurement of C-reactive protein levels | Change from baseline to 90 minutes and 120 minutes of the game.
  C-reactive protein levels will be measured on blood samples
Measurement of leukocyte counts | Change from baseline to 90 minutes and 120 minutes of the game.
  Leukocyte counts will be measured on blood samples
Measurement of Interleukin-6 levels | Change from baseline to 90 minutes and 120 minutes of the game.
  Interleukin-6 levels will be measured on blood samples
Measurement of Tumor necrosis factor - α levels | Change from baseline to 90 minutes and 120 minutes of the game.
  Tumor necrosis factor - α levels will be measured on blood samples

SECONDARY OUTCOMES:
Measurement of reactive strength index | At baseline
Measurement of blood lactate concentration | Change from baseline to 90 minutes and 120 minutes of the game.
  Lactate concentration will be measured on blood samples
Measurement of glucose concentration in blood | Change from baseline to 90 minutes and 120 minutes of the game.
  Glucose concentration will be measured on blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Prof, Principal Investigator — University of Thessaly
Locations (1):
- University of Thessaly, School of Physical Education and Sports Science, Trikala, Greece

REFERENCES:
- [Derived] Ermidis G, Mohr M, Jamurtas AZ, Draganidis D, Poulios A, Papanikolaou K, Vigh-Larsen JF, Loules G, Sovatzidis A, Nakopoulou T, Tsimeas P, Douroudos II, Papadopoulos C, Papadimas G, Rosvoglou A, Liakou C, Deli CK, Georgakouli K, Chatzinikolaou A, Krustrup P, Fatouros IG. Recovery during Successive 120-min Football Games: Results from the 120-min Placebo/Carbohydrate Randomized Controlled Trial. Med Sci Sports Exerc. 2024 Jun 1;56(6):1094-1107. doi: 10.1249/MSS.0000000000003398. Epub 2024 Jan 30. PMID 38306312
- [Derived] Mohr M, Ermidis G, Jamurtas AZ, Vigh-Larsen JF, Poulios A, Draganidis D, Papanikolaou K, Tsimeas P, Batsilas D, Loules G, Batrakoulis A, Sovatzidis A, Nielsen JL, Tzatzakis T, Deli CK, Nybo L, Krustrup P, Fatouros IG. Extended Match Time Exacerbates Fatigue and Impacts Physiological Responses in Male Soccer Players. Med Sci Sports Exerc. 2023 Jan 1;55(1):80-92. doi: 10.1249/MSS.0000000000003021. Epub 2022 Aug 12. PMID 35977104